CLINICAL TRIAL: NCT03643302
Title: Clinical Efficacy and Safety of Tran-bronchoscopy Airway Clearance and Bronchoalveolar Lavage in the Treatment of Moderate to Severe Bronchiectasis With Acute Exacerbation
Brief Title: Airway Clearance and Bronchoalveolar Lavage for Bronchiectasis Patients With Exacerbation
Status: Completed | Type: Observational
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Jin-Fu Xu, Director, Head of respiratory medicine, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: 20180717
Record Dates: First submitted 2018-08-21; First posted 2018-08-22 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Bronchiectasis Adult

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Therapy of bronchoalveolar lavage group: Patients with bronchiectasis exacerbations treat with fundamental treatment combining with the therapy of airway clearance and bronchoalveolar lavage.
  Interventions: Device: Version BF-1T26 electronic bronchoscope
- Fundamental treatment group: In the control group,fundamental treatment was adopted according to the guidelines

INTERVENTIONS:
Device: Version BF-1T26 electronic bronchoscope — Interventions involving the therapy of airway clearance and bronchoalveolar lavage by Version BF-1T26 electronic bronchoscope
  Groups: Therapy of bronchoalveolar lavage group

SUMMARY:
No study have evaluated the efficacy and safety of airway clearance therapy (ACT) and bronchoalveolar lavage (BAL) under bronchoscope for bronchiectasis.

This study aimed to evaluate the clinical efficacy and safety of tran-bronchoscopy airway clearance and bronchoalveolar lavage in the treatment of moderate to severe bronchiectasis with acute exacerbation:A randomized, prospective cohort study.

DETAILED DESCRIPTION:
The aim of this study was to evaluate the efficacy and safety of ACT combined with BAL for bronchiectasis patients with acute exacerbation through the whole study process, which will provide a high quality of evidence-based strategies for the treatment, revision and optimization of international and domestic clinical guidelines for bronchiectasis. All the participants will be required to check the various efficacy and safety indicators.

ELIGIBILITY:
Inclusion Criteria:

* Willing to join in and sign the informed consent form;
* The diagnosis of bronchiectasis need reference to the definition of "European Respiratory Society guidelines for the management of adult bronchiectasis." published by the european respiratory journal in 2017, defined by the presence of both permanent bronchial dilatation on computed tomography (CT) scanning and the clinical syndrome of cough, sputum production and/or recurrent respiratory infections;
* Pulmonary exacerbation in patients with bronchiectasis was required to meet three or more of the following key symptoms for at least 48h: Cough; Sputum volume and/or consistency; Sputum purulence; Breathlessness and/or exercise tolerance; Fatigue and/or malaise; Haemoptysis, and a clinician determines that a change in bronchiectasis treatment is required;
* According to the researchers, the subjects were willing and able to follow the protocol and were able to tolerate bronchoscopy;
* Patients with good compliance: the subject must be willing to follow the test plan requirements in the research center to complete all the assessment of the visit.

Exclusion Criteria:

* Pregnant or lactating women;
* Hypogammaglobulinemia or other autoimmune diseases;
* Clinical diagnosis of ABPA;
* Non tuberculosis mycobacteria positive 2 years before;
* Allergies or allergic to a variety of drugs;
* Poor compliance or can not cooperate judged by doctors;
* Participated in other clinical trials for nearly three months;
* The researchers considered that the subject had other circumstances that were unfit to attend;
* Suffering from a significant disease or condition outside of bronchiectasis, as judged by the researchers, may lead to subjects at risk due to participate in the study,or the disease that have an impact on the research result and the ability of subjects to participate in this study;
* Bronchoscopy contraindication;
* Patients with heart, liver and kidney, nervous system, endocrine and other systemic diseases, may not be able to adhere to the completion of the study, or will affect the research process;
* Patients who refused to sign informed consent after targeted explanation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with bronchiectasis being suffering an acute exacerbation of this disease.
Sampling Method: Non-Probability Sample
Enrollment: 189 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-03-18 (Actual)

PRIMARY OUTCOMES:
Time to the first acute exacerbation after treatment | 3 month
  The median time to first acute exacerbation after discharge.We used GraphPad Prism 6.0 Kaplan-Meier survival curve and the log-rank test to compare the differences of the primary outcome between both groups

SECONDARY OUTCOMES:
The changes of mMRC score before and after treatment | 7 days
  Modified Medical Research Centre
The changes of CAT score before and after treatment | 7 days
  COPD Assessment Test
The changes of SGRQ before and after treatment | 7 days
  St. George respiratory questionnaire
The changes of LCQ before and after treatment | 7days
  Leicester Cough Questionnaire
The changes of 6MWD before and after treatment | 1 days
  6 Minute Walking Distance

CONTACTS AND LOCATIONS:
Overall Officials: Jin-fu Xu, Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (1):
- Shanghai Pulmonary Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] McDonnell MJ, Aliberti S, Goeminne PC, Dimakou K, Zucchetti SC, Davidson J, Ward C, Laffey JG, Finch S, Pesci A, Dupont LJ, Fardon TC, Skrbic D, Obradovic D, Cowman S, Loebinger MR, Rutherford RM, De Soyza A, Chalmers JD. Multidimensional severity assessment in bronchiectasis: an analysis of seven European cohorts. Thorax. 2016 Dec;71(12):1110-1118. doi: 10.1136/thoraxjnl-2016-208481. Epub 2016 Aug 11. PMID 27516225
- [Background] Hill AT, Haworth CS, Aliberti S, Barker A, Blasi F, Boersma W, Chalmers JD, De Soyza A, Dimakou K, Elborn JS, Feldman C, Flume P, Goeminne PC, Loebinger MR, Menendez R, Morgan L, Murris M, Polverino E, Quittner A, Ringshausen FC, Tino G, Torres A, Vendrell M, Welte T, Wilson R, Wong C, O'Donnell A, Aksamit T; EMBARC/BRR definitions working group. Pulmonary exacerbation in adults with bronchiectasis: a consensus definition for clinical research. Eur Respir J. 2017 Jun 8;49(6):1700051. doi: 10.1183/13993003.00051-2017. Print 2017 Jun. PMID 28596426
- [Derived] Liu Y, Lu HW, Gu SY, Wang WW, Ge J, Jie ZJ, Jia JG, Gao ZT, Li J, Shi JY, Liang S, Cheng KB, Bai JW, Qu JM, Xu JF. Bronchoscopic airway clearance therapy for acute exacerbations of bronchiectasis. EBioMedicine. 2021 Oct;72:103587. doi: 10.1016/j.ebiom.2021.103587. Epub 2021 Sep 16. PMID 34537448